CLINICAL TRIAL: NCT04753944
Title: Probiotics Therapy: a New Approach to Therapy of Mood Disorders in Perimenopausal Women
Brief Title: Probiotics Therapy of Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Ewa Stachowska, Professor, head of Department of Human Nutrition and Metabolimics. PhD, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pomeranian Medical Univeristy
Record Dates: First submitted 2020-05-07; First posted 2021-02-15 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: probiotics; mood; depressive; therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Intervention, randomized, double-blind, using placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and investigators enrolling participants could not foresee assignment because to conceal allocation equentially numbered probiotic containers of identical appearance was used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Patients will be introduced for 5 weeks with probiotic therapy (in the study group). They will take Ecologic®Barrier (Winclove Probiotics BV, Amsterdam, The Netherlands), consisting of Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19 and Lactococcus lactis W58. The probiotic dose is going to be 4 capsules daily (one capsule contains 500 million CFUs of living probiotic strains). The treatment will be administered two times a day, during breakfast and supper. The probiotic formula will be Provided by polish distributor of Winclove products, namely Sanprobi sp. z o. o. sp. k
  Interventions: Dietary Supplement: Active Comparator: Probiotic
- Placebo group (Placebo Comparator): Patients will be introduced for 5 weeks with placebo that consist of maize starch, maltodextrins and vegetable protein. The placebo dose is going to be 4 capsules daily (one capsule). The treatment will be administered two times a day, during breakfast and supper.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Active Comparator: Probiotic — The evaluation of the influence of a probiotics therapy on mood improvement and the reduction of depressive symptoms in women in the perimenopausal age group.
  Other Names: Probiotic Ecologic®Barrier (Winclove Probiotics BV)
  Arms: Probiotic group
Dietary Supplement: Placebo group — Patients will be introduced for 5 weeks with placebo consisting of starch, maltodextrins and vegetable protein. The placebo dose is going to be 4 capsules daily. The treatment will be administered two times a day, during breakfast and supper.
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
The evaluation of the influence of a probiotics therapy on mood improvement and the reduction of depressive symptoms in women in the perimenopausal age group.

DETAILED DESCRIPTION:
The aim: The evaluation of the influence of a probiotics therapy on mood improvement and the reduction of depressive symptoms in women in the perimenopausal age group.

The study hypothesis: By using periodic probiotics therapy it is possible to positively influence the mood of women with depressive syndromes. These efforts focus on the improvement of the functioning of the gut barrier and gut-brain axis. In practice, such activities should lead to the reduction in the dysfunction of the barrier, the reduction of endotoxemia and the concentration of neurotoxic metabolites of tryptophan (in blood) with the simultaneous increase in the content of butyric acid that has a neuroprotective effect.

The of the trial: intervention, cohort, randomized, double-blind, using placebo. A multi-strain probiotic will also be provided ( Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19 and Lactococcus lactis W58 or maize starch, maltodextrins and vegetable protein/placebo).

The applied method of study:

1. a controlled dietary intervention that includes probiotics therapy; the verification of the past nutritional pattern (the Food Frequency Questionnaire); anthropometric measurements;
2. psychiatric studies: the evaluation of sleep disorders (the Athens insomnia scale) and mood (the Beck scale), and the worsening of depression (the Hamilton scale);
3. biochemical studies: the content of short chain fatty acids (in the stool);
4. cytometric studies (B-type lymphocytes' panel, T-type lymphocytes' panel, regulatory T cells' panel);
5. genetic (the microbiome of bacteria in the stool, pyrosequencing);
6. chromatographic (the derivatives of tryptophan e.g., kynurenine, anthranilic acid, kynureic acid, 3-hydroxykynurenine, 5-hydroxytryptophan, serotonin).

Currently, there is an urgent problem to develop recommendations regarding the nutrition and probiotics therapy that could complement the therapy of women with mood disorders. If the achieved results confirm the study hypothesis, it will be possible to:

1. better understand the pathomechanism of mood disorders in the perimenopausal period;
2. develop a holistic strategy for depressive disorders in women in the menopause period.

ELIGIBILITY:
Inclusion Criteria:

* must presence of mood disorders confirmed by Beck scale (more than 10 points)
* must be able to swallow tablets

Exclusion Criteria:

* individuals that had prescribed antibiotics, proton pump inhibitors, or probiotics in the 6 months preceding the study (eg. inflammatory bowel syndrome)
* circulatory disorders patients
* diagnosed coagulopathies,
* diagnosed respiratory disease
* inflammatory bowel disease patients
* addicted to alcohol
* addicted to psychoactive substances,

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Perimenopausal women are qualified for examinations (based on medical and hormonal examination) at the Clinic of Gynecology, Endocrinology and Gynecology PUM.
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Dietary intervention | 5 weeks
  The verification of the past nutritional pattern (will be asses by Food Freguency Questionnarie). The indicate frequency of food consumption, respondents could choose one of six categories (next converted by researcher into daily frequency): never or very rarely (0 times/day), once a month or less (0.025 times/day), several times a month (0.1 times/day), several times a week (0.571 times/day), daily (1 time/day), or a few times a day (2 times/day)
Anthropometric measurements | 5 weeks
  The verification of body mass during the study will be asses by body mass index (BMI). In order of this, we will measure the height (outcome in cm). BMI will be calculated by dividing body weight (in kilograms) by height squared (in meters).i Finally BMI will be presented in kg/m2.
Depression intensity mesurements | 5 weeks
  Depression intensity will be asses by the Hamilton Rating Scale for Depression (HRSD).Unit HRSD ( 0-7 not depressed, 8-13 mild depression; 14-18 moderate depression (mild); 19-22 moderate depression; > 23 severe depression)
The biochemical changes in stool | 5 weeks
  Observation of biochemical changes short fatty acids (SCFAs) concentration before and after the intervention (SCFA in ng/ml)
The cytometric studies | 5 weeks
  Observation of a change in Mean Fluorescence Intensity (FSC) of lymphocytes B and regulatory T cells before and after intervention in flow cytometry. Assessments by median: midpoint of the population (middle channel)).
The stool microbiota changes | 5 weeks
  Changes in gut microbiota composition and metabolism (16 SrRNA bacterial genomic, bacterial metabolites) at enrollment and at the end-point ( gut microbiota will be asses in Operational taxonomic units (OTUs))
Insomnia studies | 3 months
  Assessments using unique measurements Athens insomnia scale ( 0 to < 6 means no insomnia; more than 6 points indicated diagnosis of insomnia)
The Kynureine Pathway | 3 months
  The changes in the tryptophan pathway derivatives before and after intervention will be measured. ( we assess metabolites of kynurenine pathway e.g. 5 HT, HIAA, KYN will be asses by HPLC (in ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Samochowiec, prof, MD, Study Director — Pomeranian Medical University in Sczecin
Locations (1):
- Pomeranian Medical University, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No